CLINICAL TRIAL: NCT02265536
Title: Phase 1 Study to Identify the Immunomodulatory Activity of LY3022855 (IMC-CS4) in Patients With Advanced, Refractory Breast or Prostate Cancer
Brief Title: A Study of LY3022855 In Participants With Breast or Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15441; I5F-MC-JSCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-09-24; First posted 2014-10-16 (Estimated); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — LY3022855

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY3022855 1.25 mg/kg Q2W (Experimental): 1.25 milligram per kilogram (mg/kg) LY3022855 administered intravenously (IV), once every two weeks (Q2W). Treatment is 6 week cycle. Participants may receive multiple cycles if they are deriving clinical benefit.
  Interventions: Drug: LY3022855
- LY3022855 1.0 mg/kg WK1_2_4_5 (Experimental): 1.0 mg/kg LY3022855 administered IV on Weeks 1, 2, 4, and 5 of a 6-week cycle. Participants may receive multiple cycles if they are deriving clinical benefit.
  Interventions: Drug: LY3022855
- LY3022855 100 mg Q2W (Experimental): 100 mg of LY3022855 administered IV once every two weeks of a 6-week cycle. Participants may receive multiple cycles if they are deriving clinical benefit.
  Interventions: Drug: LY3022855
- LY3022855 100 mg QW (Experimental): 100 mg of LY3022855 administered IV. once a week (QW) of a 6-week cycle. Participants may receive multiple cycles if they are deriving clinical benefit.
  Interventions: Drug: LY3022855

INTERVENTIONS:
Drug: LY3022855 — Administered IV
  Other Names: IMC-CS4

SUMMARY:
The main purpose of this study is to learn more about how the investigational drug, LY3022855, affects the immune system in participants with advanced breast or prostate cancer that has not responded to other treatments. Treatment may last up to 6 cycles (cycle = 6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of advanced, refractory breast or prostate cancer that is evaluable by radiologic testing. Participants must have experienced tumor progression on or treatment intolerance to at least one prior therapy and have declined or are ineligible for a standard treatment.
* For participants with metastatic castrate-resistant prostate cancer only:

  * Must continue ongoing androgen deprivation therapy with castrate levels of serum testosterone <50 nanogram/deciliter (ng/dL) determined within 4 weeks prior to starting treatment
  * If receiving an antiandrogen as part of first-line hormonal therapy, must have shown progression of disease off the antiandrogen prior to enrollment
  * Must be willing to continue androgen deprivation therapy while on study, if no prior orchiectomy
  * Must meet at least 1 of the following 3 criteria for progressive metastatic disease, according to Prostate Cancer Working Group 2 (PCWG2) criteria:

    * A rise in prostate-specific antigen (minimal value 2 ng/milliliter (mL); ≥3 consecutive rising values)
    * ≥2 new metastases on transaxial imaging or radionuclide bone scan
    * Soft tissue progression
  * Replacement hormone therapy initiated before study entry is permitted
  * For participants with breast cancer only:

    * May continue ongoing antiestrogen therapy
    * Replacement hormone therapy initiated before study entry is permitted
    * May continue ongoing trastuzumab therapy
* Have adequate organ and hematologic function, including: Hepatic: Bilirubin ≤1.5 × the upper limit of normal (ULN), and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 × ULN. For participants with tumor involvement of the liver, AST and ALT ≤5.0 × ULN are acceptable. For participants with tumor involvement of the bone, alkaline phosphatase ≤5.0 × ULN is acceptable. Renal: Serum creatinine ≤2.0 × ULN. Absolute neutrophil count (ANC) ≥1.0 × 10^9/liter (L). Hemoglobin ≥9 grams per deciliter (5.58 millimoles per liter). Platelets ≥90 × 10^9/L.
* Have Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Have discontinued all disease-modifying therapy for the primary cancer >28 days prior to initiation of study treatment. In addition, clinically significant toxicities associated with any prior therapy for the primary cancer, including investigational treatments, have resolved or stabilized to Grade ≤1 toxicity >28 days prior to initiation of study treatment with the exception of neuropathy, which must have resolved to Grade ≤2. Continuation of a stable dose (minimum of 28 days prior to study entry) of denosumab or bisphosphonate is permitted on study.
* Willing and able to comply with study procedures including 1 baseline and 1 posttreatment tumor biopsy procedure.
* Male participants: Agree to use a reliable method of birth control and to not donate sperm during the study and for at least 12 weeks following last dose of study drug or country requirements, whichever is longer.
* Female participants: Are women of child-bearing potential who test negative for pregnancy within 7 days prior to enrollment based on a urine or serum pregnancy test and agree to use a reliable method of birth control during the study and for 12 weeks following the last dose of the study drug and also must not be breastfeeding, OR are postmenopausal women.
* Have an estimated life expectancy that, in the judgment of the investigator, will permit the patient to complete 1 cycle of treatment.
* May have received treatment with an investigational product or non-approved use of a drug (other than the study drug used in this study) or device for non-cancer indications; however, not within 28 days prior to the initial dose of study drug.

Exclusion Criteria:

* Have received treatment within 28 days prior to the initial dose of study drug with an investigational product or non-approved use of a drug or device (other than the study drug/device used in this study) for non-cancer indications or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have serious preexisting medical conditions (left to the discretion of the investigator).
* Have symptomatic central nervous system (CNS) malignancy or metastasis.
* Have an active fungal, bacterial, and/or known viral infection, including human immunodeficiency virus (HIV) or viral (B or C) hepatitis.
* Have any of the following cardiovascular conditions:

  * Symptomatic coronary artery disease currently or within the past 6 months,
  * Have a second active primary malignancy that, in the judgment of the investigator or sponsor, may affect the interpretation of the results.
  * Confirmed left ventricular ejection fraction ≤50% or any cardiac insufficiency > New York Heart Association (NYHA) class II currently or within the past 6 months,
  * Uncontrolled hypertension (>170/100 millimeter of mercury [mm Hg]) currently or within the past 7 days, or
  * Serious cardiac arrhythmia (well-controlled atrial fibrillation is permitted) currently or within the past 6 months.
* Have a second active primary malignancy that, in the judgment of the investigator or sponsor, may affect the interpretation of the results.
* Are unwilling or unable to participate in tumor biopsies.
* Have corrected QT interval of >500 millisecond (msec) on screening electrocardiogram (ECG).
* Have received treatment with agents specifically targeting colony stimulating factor 1 (CSF-1) or CSF-1R, including imatinib, nilotinib, and sunitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Autio KA, Klebanoff CA, Schaer D, Kauh JSW, Slovin SF, Adamow M, Blinder VS, Brahmachary M, Carlsen M, Comen E, Danila DC, Doman TN, Durack JC, Fox JJ, Gluskin JS, Hoffman DM, Kang S, Kang P, Landa J, McAndrew PF, Modi S, Morris MJ, Novosiadly R, Rathkopf DE, Sanford R, Chapman SC, Tate CM, Yu D, Wong P, McArthur HL. Immunomodulatory Activity of a Colony-stimulating Factor-1 Receptor Inhibitor in Patients with Advanced Refractory Breast or Prostate Cancer: A Phase I Study. Clin Cancer Res. 2020 Nov 1;26(21):5609-5620. doi: 10.1158/1078-0432.CCR-20-0855. Epub 2020 Aug 26. PMID 32847933
- See also: A Study of LY3022855 In Participants With Breast or Prostate Cancer — https://www.lillytrialguide.com/en-US/studies/breast-cancer/JSCB#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died from any cause or disease progression and participants who were alive and on study (either on study treatment or in long term follow-up) at study conclusion.
Groups:
- LY3022855 - 1.25 mg/kg Q2W Breast Cancer: Participants received 1.25 milligram per kilogram (mg/kg) of LY3022855 administered intravenously (IV) once every two weeks (Q2W) of a 6-week cycle.
- LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer; LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer: Participants received 1.0 mg/kg of LY3022855 administered IV on Weeks
  1, 2, 4, and 5 of a 6-week cycle.
- LY3022855 - 100 mg Q2W Breast Cancer: Participants received 100 mg of LY3022855 administered IV once every two weeks of a 6-week cycle.
- LY3022855 - 100 mg QW Breast Cancer: Participants received 100 mg of LY3022855 administered IV once weekly (QW) of a 6-week cycle.
- LY3022855 - 1.25 mg/kg Q2W Prostate Cancer: Participants received 1.25 mg/kg of LY3022855 administered IV once every two weeks of a 6-week cycle.
Period: Overall Study
Arm/Group | LY3022855 - 1.25 mg/kg Q2W Breast Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer | LY3022855 - 100 mg Q2W Breast Cancer | LY3022855 - 100 mg QW Breast Cancer | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer
Started | 6 | 5 | 5 | 6 | 8 | 4
Received at Least 1 Dose of Study Drug | 6 | 5 | 5 | 6 | 8 | 4
Completed | 5 | 2 | 5 | 6 | 5 | 4
Not Completed | 1 | 3 | 0 | 0 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- LY3022855 - 1.25 mg/kg Q2W Breast Cancer; LY3022855 - 1.25 mg/kg Q2W Prostate Cancer: Participants received 1.25 mg/kg of LY3022855 administered IV once every two weeks of a 6-week cycle.
- LY3022855 - 100 mg QW Breast Cancer: Participants received 100 mg of LY3022855 administered IV once weekly of a 6-week cycle.
- Total: Total of all reporting groups
Arm/Group | LY3022855 - 1.25 mg/kg Q2W Breast Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer | LY3022855 - 100 mg Q2W Breast Cancer | LY3022855 - 100 mg QW Breast Cancer | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer | Total
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 8 | 4 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (16.6) | 55.4 (11.8) | 54.8 (10.7) | 58.3 (16.1) | 69.8 (8.3) | 71.0 (9.2) | 60.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 3 | 6 | 0 | 0 | 20
  Male | 0 | 0 | 2 | 0 | 8 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 5 | 5 | 6 | 8 | 4 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 5 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 2 | 4
  White | 4 | 5 | 3 | 0 | 8 | 2 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 5 | 6 | 8 | 4 | 34
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram/Meter^2 (kg/m^2)] | 27.3 (6.0) | 26.5 (6.0) | 24.2 (4.8) | 25.1 (4.5) | 27.8 (3.4) | 28.6 (6.2) | 26.6 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Peripheral Blood Immune Cell (PBIC) Subsets
Description: The immunomodulatory activity of the drug was documented by examining markers that include, but are not limited to: Live-Dead, Cluster of Differentiation 3 (CD3), CD4, CD8, CD14, CD16, Foxhead Box p3 (FoxP3), PD-1, Ki-67, Cytotoxic T-Lymphocyte Antigen 4 (CTLA-4), Human Leukocyte Antigen-D-relate (HLA-DR), T-cell immunoglobulin and mucin-3 (TIM-3), lymphocyte-activation gene 3 (LAG-3), and Inducible T-cell COStimulator (ICOS). The expression of these markers was quantified by flow cytometric analysis with an antibody panel.
Time Frame: Baseline to Day 8 after 1st dose
Population: All enrolled participants who received at least one dose of study drug and have baseline and post baseline data for peripheral blood immune cell subsets.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | LY3022855 - 1.25 mg/kg Q2W Breast Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer | LY3022855 - 100 mg Q2W Breast Cancer | LY3022855 - 100 mg QW Breast Cancer | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 8 | 4
Percent Change
  C14_HLA_DR_%: number analyzed (Participants) | 5 | 3 | 2 | 2 | 8 | 2
  C14_HLA_DR_% | -10.31 [-39.58 to -9.05] | 5.12 [1.54 to 26.3] | -16.39 [-21.73 to -11.05] | -26.76 [-28.66 to -24.87] | -11.77 [-19.97 to -1.71] | -11.72 [-15.71 to -7.73]
  LIVE_CELL_Count (CNT): number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  LIVE_CELL_Count (CNT) | -9.85 [-13.45 to -3.18] | -20.08 [-26.37 to -1.67] | -12.82 [-39.07 to 4.13] | 1.23 [-7.11 to 10.71] | 0.43 [-10.33 to 7.02] | -3.48 [-3.82 to -3.28]
  CD3_CNT: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CD3_CNT | -10.53 [-24.82 to -0.59] | 39.23 [-8.69 to 77.95] | 1.92 [-20.92 to 16.58] | -19.27 [-27.82 to 17.61] | 12.35 [-3.29 to 19.26] | -2.35 [-10.44 to 8.31]
  CD3_LIVE_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CD3_LIVE_% | -3.54 [-17.62 to 5.09] | 16.63 [-11.76 to 33.86] | 20.32 [13.89 to 36.08] | -5.33 [-8.5 to 4.87] | 8.11 [-4.29 to 20.15] | -5.11 [-10.76 to -1.17]
  CD4_CD3_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CD4_CD3_% | 1.81 [-2.97 to 9.84] | 3.18 [-0.35 to 5.16] | -3.01 [-4.49 to 0.29] | -0.15 [-14.67 to 10.5] | 0.41 [-1.24 to 1.67] | 7.34 [0 to 10.65]
  CD4_CNT: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CD4_CNT | -13.02 [-22.31 to 2.58] | 43.43 [-6.95 to 86.22] | 2.87 [-17.63 to 13.04] | -18.79 [-38.14 to 17.61] | 11.31 [-2.75 to 18.02] | 4.65 [-1.27 to 7.45]
  CD8_CD3_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CD8_CD3_% | -4.02 [-10.44 to 4.76] | -4.5 [-9.56 to 3.45] | 1.96 [-7.73 to 8.53] | 28.25 [13.74 to 37.77] | 0 [-8.71 to 4.82] | -9.91 [-16.93 to 11.77]
  CD8_CD4_RATIO: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CD8_CD4_RATIO | -5.53 [-18.34 to 7.93] | -7.44 [-13.77 to 4.7] | 0.01 [-10.97 to 11.13] | 32.87 [21 to 49.28] | 0.4 [-11.34 to 5.67] | -16.13 [-24.67 to 14.1]
  CD8_CNT: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CD8_CNT | -6.41 [-28.35 to -0.63] | 29.87 [-11.54 to 61.92] | 4.58 [-25.47 to 26.47] | -9.9 [-12.59 to 51.2] | 13.01 [-10.94 to 18.46] | -12.32 [-25.17 to 23.42]
  CD8_FOXP3_RATIO: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CD8_FOXP3_RATIO | -10.61 [-18.7 to -1.07] | -17.56 [-19.76 to 3.97] | 28.48 [18.76 to 38.75] | 123.96 [10.17 to 230.5] | -4.12 [-21.58 to 11.66] | -0.64 [-4.91 to 15.96]
  CTLA4_CD4_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CTLA4_CD4_% | 4.14 [-6.63 to 13.34] | 18.49 [-3.27 to 36.61] | -26.26 [-37 to -15.26] | 2.18 [-30.98 to 31.16] | 31.67 [1.37 to 44.97] | 3.59 [-9.12 to 13.74]
  CTLA4_CD8_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  CTLA4_CD8_% | -7.34 [-16.22 to 9.76] | 19.43 [-56.63 to 97.71] | -21.33 [-25.18 to -3.45] | -11 [-50.03 to 56.66] | 7.48 [-4.19 to 35.05] | -10.32 [-24.03 to 47.92]
  FOXP3_CD4_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  FOXP3_CD4_% | 26.31 [-2 to 30.37] | 2.39 [-11.76 to 14.97] | -21.12 [-39.09 to -1.69] | -33.46 [-45.31 to -13.45] | 13.51 [-11.69 to 18.56] | -7.74 [-20.29 to 0.38]
  FOXP3_CD8_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  FOXP3_CD8_% | 35.94 [21.09 to 39.73] | -7.17 [-32.96 to 2.97] | -48.43 [-49.7 to -46.03] | -33.81 [-69.36 to 2.12] | 20.36 [12.26 to 58.96] | 52.01 [8.22 to 84.24]
  FOXP3_CNT: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  FOXP3_CNT | -7.43 [-22.89 to 16.7] | 63.34 [6.29 to 97.2] | -18.38 [-51.04 to 11.19] | -51.05 [-72.49 to -11.58] | 2.37 [-8.31 to 29.16] | -3.16 [-20.42 to 8.25]
  ICOS_CD4_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  ICOS_CD4_% | -5.72 [-12.92 to -2.46] | 0.77 [-5.46 to 25.56] | -14.6 [-24.04 to -0.44] | 17.69 [-4.46 to 32.57] | 30.4 [-0.37 to 46.77] | 17.76 [2.74 to 48.27]
  ICOS_CD8_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  ICOS_CD8_% | 3.75 [-19.71 to 8.05] | 17.18 [-8.75 to 31.03] | -30 [-38.78 to -7.52] | -18.81 [-35.45 to 10.09] | 9.08 [-28.61 to 23.41] | -25.12 [-26.37 to -23.36]
  KI67_CD4_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  KI67_CD4_% | -17.44 [-24.98 to -7.28] | 70.56 [19.8 to 101.12] | -30.52 [-36.48 to -26.81] | -6.57 [-51.21 to 63.09] | 0.19 [-10.34 to 73.56] | 8.18 [-9.64 to 62.58]
  KI67_CD8_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  KI67_CD8_% | -27.13 [-54.17 to 0.66] | 17.47 [-12.49 to 60.93] | -15.46 [-27.25 to 0.17] | -7.75 [-54.51 to 70.84] | -6.48 [-20.64 to 63.7] | -3.75 [-15.92 to 64.4]
  LAG3_CD4_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  LAG3_CD4_% | 87.25 [44.31 to 106.7] | -18.38 [-42.96 to 10.36] | -15.67 [-38.96 to 31.72] | 10.35 [-14.07 to 44.06] | 40.36 [17.91 to 74.15] | 9.74 [9.68 to 16.55]
  LAG3_CD8_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  LAG3_CD8_% | 59.83 [9.63 to 101.28] | -24.98 [-31.79 to -13.65] | 3.48 [-26.54 to 42.81] | 69.63 [45.48 to 98.24] | 7.87 [-2.89 to 58.77] | 80.24 [23.83 to 81.04]
  PD1_CD4_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  PD1_CD4_% | -6.58 [-12.48 to 3.18] | 15.71 [11.46 to 22.05] | -5.25 [-12.67 to 4.02] | 19.18 [6.39 to 26.88] | -13.58 [-28.27 to 10.3] | 4.14 [-3.18 to 50.31]
  PD1_CD8_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  PD1_CD8_% | -14.49 [-18.09 to -8.19] | 8.32 [-9.13 to 25.82] | -2.49 [-17.22 to 21.96] | 20.59 [9.1 to 24.82] | -11.85 [-20 to 20.32] | -2.2 [-15.81 to 35.46]
  TIM3_CD4_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  TIM3_CD4_% | -36.63 [-38.64 to -16.56] | -29.87 [-30.86 to -0.59] | -15.45 [-21.9 to -8.64] | -21.93 [-40.21 to -7.64] | -12.12 [-19.61 to -0.92] | -18.49 [-25.07 to -12.18]
  TIM3_CD8_%: number analyzed (Participants) | 6 | 4 | 4 | 4 | 8 | 3
  TIM3_CD8_% | 1.53 [-4.03 to 24.46] | 1.69 [-12.29 to 16.18] | 6.18 [-13.76 to 25.2] | -16.65 [-21.76 to -4.47] | 0.7 [-20.5 to 31.25] | -33.08 [-43.49 to -30.02]
  CD14DIM_CD16BR_%: number analyzed (Participants) | 5 | 3 | 4 | 4 | 7 | 3
  CD14DIM_CD16BR_% | -95.12 [-96.15 to 72.73] | 12.24 [-40.59 to 25.44] | -60.59 [-82.14 to -10.19] | -95.09 [-96.81 to -91.77] | -88.73 [-94.44 to -75.81] | -92.73 [-95.2 to -52.61]

2. Primary Outcome: Percentage Change From Baseline in Serum Cytokines
Description: The immunomodulatory activity of the drug was measured in participants with advanced, refractory breast or prostate cancers using serum cytokines. Serum cytokine levels was determined by MSD multiplex cytokine immunoassay technology or ELISA, and that may include but not be limited to Interleukin 6 (IL-6), IL-8, IL-10 and Tumor necrosis factor (TNF-α).
Time Frame: Baseline to Day 8 after 1st dose
Population: All enrolled participants who received at least one dose of study drug and have baseline and post baseline data for Serum Cytokines.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | LY3022855 - 1.25 mg/kg Q2W Breast Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer | LY3022855 - 100 mg Q2W Breast Cancer | LY3022855 - 100 mg QW Breast Cancer | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 8 | 4
Percent Change
  TNF-α: number analyzed (Participants) | 5 | 4 | 1 | 3 | 5 | 0
  TNF-α | -14.51 [-19.84 to 81.88] | 48.28 [16.56 to 61.5] | 416.95 [416.95 to 416.95] | 3.51 [-21.14 to 14.91] | 6.1 [-14.11 to 61.5] |
  IL-8: number analyzed (Participants) | 6 | 5 | 5 | 6 | 8 | 3
  IL-8 | 24.53 [18.82 to 7901] | 62.84 [-38.78 to 189.47] | 1956.66 [1108.74 to 2804.58] | -19.97 [-41.55 to 435.42] | 67.42 [29.18 to 122.35] | -7.62 [-51.64 to 57.42]
  IL-6: number analyzed (Participants) | 5 | 4 | 2 | 3 | 8 | 2
  IL-6 | 18.13 [-38.15 to 35.79] | 35.76 [-9.31 to 72.08] | 1956.66 [1108.74 to 2804.58] | -19.97 [-41.55 to 435.42] | 67.42 [29.18 to 122.35] | -7.62 [-51.64 to 57.42]
  IL-10: number analyzed (Participants) | 5 | 4 | 0 | 0 | 4 | 0
  IL-10 | 83.3 [45.6 to 94.11] | 12.69 [-41.7 to 95.05] |  |  | 174.75 [139.08 to 191.88] |

3. Primary Outcome: Serum Cytokine Levels
Description: The immunomodulatory activity of the drug was measured in participants with advanced, refractory breast or prostate cancers using serum cytokines. Serum cytokines will be determined by MSD multiplex cytokine immunoassay or ELISA. The markers to be measured using these technologies include, but are not limited to: CSF-1, IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, IL-34, and TNF-α.
Time Frame: Day 8
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: nanograms per liter (ng/L)
Arm/Group | LY3022855 - 1.25 mg/kg Q2W Breast Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer | LY3022855 - 100 mg Q2W Breast Cancer | LY3022855 - 100 mg QW Breast Cancer | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 7 | 4
nanograms per liter (ng/L)
  CSF-1 | 308460 [182347.5 to 358665] | 23564.3 [511.4 to 70952.5] | 290520 [792.8 to 328780] | 470350 [335340 to 472700] | 235950 [67192 to 247580] | 159550 [81224.5 to 211830]
  IL-34 | 670.6 [425.75 to 766.08] | 137.56 [62.5 to 257.73] | 498.89 [62.5 to 637.28] | 447.11 [357.36 to 737.66] | 392.54 [145.57 to 517.92] | 123.44 [106.27 to 167.87]

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve of LY3022855
Description: Area under the concentration versus time curve from time zero to tau (τ) of LY3022855 (AUC[0- τ]), where tau is dosing interval of (0-14 days).
Time Frame: 0, 1, 4, 24, 48, 72 and 168 hours post dose on Day 1 and Day 29
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data for AUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms/mL
Groups:
- LY3022855 - 1.25 mg/kg Q2W: Participants received 1.25 mg/kg of LY3022855 administered IV once every two weeks of a 6-week cycle.
- LY3022855 - 1.0 mg/kg WK1_2_4_5: Participants received 1.0 mg/kg of LY3022855 administered IV on weeks 1, 2, 4, and 5 of a 6-week cycle.
- LY3022855 - 100 mg Q2W: Participants received 100 mg of LY3022855 administered IV once every two weeks of a 6-week cycle.
- LY3022855 - 100 mg QW: Participants received 100 mg of LY3022855 administered IV once weekly of a 6-week cycle.
Arm/Group | LY3022855 - 1.25 mg/kg Q2W | LY3022855 - 1.0 mg/kg WK1_2_4_5 | LY3022855 - 100 mg Q2W | LY3022855 - 100 mg QW
Number analyzed (Participants) | 6 | 5 | 4 | 2
hours*micrograms/mL
  Day 1 | 1950 (35) | 1030 (38) | 4310 (14) | 2350 (31)
  Day 29: number analyzed (Participants) | 6 | 0 | 0 | 0
  Day 29 | 2260 (61) |  |  |

5. Secondary Outcome: Percentage of Participants With a Best Overall Disease Control Response (Disease Control Rate)
Description: Disease control rate is the percentage of participants with a confirmed CR, PR or SD, as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1. CR is the disappearance of all target and non-target lesions; PR is a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesion; SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Disease control rate is calculated as a total number of participants with CR or PR or SD divided by the total number of participants treated, then multiplied by 100.
Time Frame: Baseline up to 6 cycles (cycle = 6 weeks)
Population: All enrolled participants who received at least one dose of study drug and have baseline and post-baseline data for disease control rate.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LY3022855 - 1.25 mg/kg Q2W Breast Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer | LY3022855 - 100 mg Q2W Breast Cancer | LY3022855 - 100 mg QW Breast Cancer | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 8 | 4
Percentage of Participants | 50 [15.3 to 84.7] | 0 [0 to 0] | 20 [1 to 65.7] | 16.7 [0.9 to 58.2] | 37.5 [11.1 to 71.1] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Up To 133 Weeks
Description: All enrolled participants who received at least 1 dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | LY3022855 - 1.25 mg/kg Q2W Breast Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer | LY3022855 - 100 mg Q2W Breast Cancer | LY3022855 - 100 mg QW Breast Cancer | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/5 | 1/5 | 1/6 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/5 | 1/5 | 1/6 | 4/8 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 5/5 | 6/6 | 8/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3022855 - 1.25 mg/kg Q2W Breast Cancer (N=6) | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer (N=5) | LY3022855 - 100 mg Q2W Breast Cancer (N=5) | LY3022855 - 100 mg QW Breast Cancer (N=6) | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer (N=8) | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease complication (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY3022855 - 1.25 mg/kg Q2W Breast Cancer (N=6) | LY3022855 - 1.0 mg/kg WK1_2_4_5 Breast Cancer (N=5) | LY3022855 - 100 mg Q2W Breast Cancer (N=5) | LY3022855 - 100 mg QW Breast Cancer (N=6) | LY3022855 - 1.25 mg/kg Q2W Prostate Cancer (N=8) | LY3022855 - 1.0 mg/kg WK1_2_4_5 Prostate Cancer (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (4) | 2 (2) | 1 (1) | 2 (2) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (1) | 2 (2) | 5 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (2) | 3 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (6) | 3 (3) | 2 (2) | 3 (4) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (5) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 3 (3) | 3 (4) | 3 (4) | 7 (10) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2) | 1 (5) | 0 (0) | 4 (5) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 1 (3) | 2 (5) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (8) | 0 (0) | 2 (3) | 2 (4) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (4) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (5) | 0 (0) | 2 (7) | 3 (6) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (5) | 1 (1) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 0 (0) | 3 (7) | 2 (2) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0/0 (0) | 0/0 (0) | 0/2 (0) | 0/0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (6) | 1 (1) | 4 (5) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Breast disorder (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/3 (0) | 0 (0) | 0/0 (0) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT02265536/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT02265536/SAP_001.pdf